CLINICAL TRIAL: NCT06885489
Title: The Effect of Acceptance and Commitment Therapy-Based Intervention on Depression, Anxiety, Stress and Psychological Well-Being Levels in University Students
Brief Title: The Effect of Acceptance and Commitment Therapy-Based Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ceylan Aksoy, Principal Investigator, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: E-95531838-050.99-124695
Record Dates: First submitted 2025-03-12; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Mental Disorder; Depression Disorders; Stress; Anxiety; Acceptance and Commitment Therapy; Psychological Well-being
MeSH Terms: conditions — Mental Disorders; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACT Intervention Group (Experimental): The group receiving Acceptance and Commitment Therapy (ACT)-based intervention.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT) based psychoeducation program
- Control Group (No Intervention): No intervention group

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) based psychoeducation program — This study implements an ACT-based psychological intervention designed to enhance psychological well-being and reduce depression, anxiety, and stress among university students. The intervention consists of structured sessions focusing on psychological flexibility, mindfulness, acceptance, and value-driven actions. Participants engage in experiential exercises, cognitive defusion techniques, and behavioral commitment strategies. The intervention is delivered over 8 weeks, with weekly sessions lasting approximately 40 minutes. The sessions are conducted in groups by trained professionals.
  Arms: ACT Intervention Group

SUMMARY:
Mental health is essential for students' emotional, cognitive, and social well-being. University life presents significant academic, social, and financial challenges, leading to increased stress, anxiety, and depression. These psychological difficulties negatively impact students' academic performance, relationships, and overall quality of life. Despite these challenges, many students avoid seeking professional help.

Acceptance and Commitment Therapy (ACT) is an effective approach that enhances psychological resilience and helps individuals cope with stress, anxiety, and depression. Instead of changing negative thoughts, ACT fosters psychological flexibility, encouraging individuals to develop a healthier relationship with them. Research supports ACT's effectiveness in reducing psychological distress, improving emotional regulation, and enhancing life satisfaction

ELIGIBILITY:
Inclusion Criteria:

* ust be currently enrolled as a full-time student at a university.

Exclusion Criteria:

* Individuals with significant cognitive impairments or those unable to understand the study procedures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scale (DASS-21) | 8 week
  DASS-21 is the short version of the Depression, Anxiety and Stress Scale-42 (DASS-42) developed by Lovibond and Lovibond. The Turkish adaptation of the scale was made by Sarıçam. The 4-point Likert-type scale includes a total of 21 items consisting of three sub-dimensions: depression, anxiety and stress. In the normal sample, test-retest reliability coefficients were found to be r=0.68 for depression, r=0.66 for anxiety and r=0.61 for stress. An individual's score of 5 and above on the depression sub-scale, 4 and above on the anxiety sub-scale and 8 and above on the stress sub-scale is interpreted as indicating the relevant psychological problem.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk Üniversitesi, Erzurum, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No